CLINICAL TRIAL: NCT06726356
Title: Efficacy and Safety of Bronchoalveolar Lavage with Acetylcysteine in the Treatment of Bronchiectasis with Infection in Adults: a Multicentre, Blinded, Randomised Controlled Study.
Brief Title: Value of Bronchoalveolar Lavage with Acetylcysteine in the Treatment of Bronchiectasis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Collaborators: Shenzhen Third People's Hospital (Other); Anhui Chest Hospital (Other); Ninghai First Hospital (Unknown); Jingzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-R036-01
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bronchiectasis with Acute Exacerbation
Keywords: bronchiectasis; acetylcysteine; bronchoalveolar lavage; Bronchoscopic airway clearance therapy
MeSH Terms: conditions — Bronchiectasis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Intervention Model Description: Control group A (conventional clinical treatment), Control group B (application of saline bronchoalveolar lavage based on conventional clinical treatment), and group C (application of bronchoscopic acetylcysteine combined with saline alveolar lavage based on conventional clinical treatment), were randomly selected into the groups according to a predefined sequence of randomisation tables prior to the operation due to the nature of the intervention.
Who Masked: Participant
Masking Description: Subjects were blinded. Study personnel responsible for assessing patients' symptom scores and recording information on acute exacerbations were blinded whenever possible. The bronchoscopy operator responsible for giving bronchoalveolar lavage treatment and the person in charge of the patient's bed were not blinded. To avoid subjective bias on the part of the assessor, non-blind people should not disclose blinded information to the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (No Intervention): based on conventional clinical treatment including anti-infective and expectorant therapy.
- Group B (Other): Bronchoalveolar lavage with saline on the basis of conventional clinical treatment, with a volume of 90 ml per target lung lobe, up to a maximum of 2 lobes, and a total volume of up to 180 ml.
  Interventions: Procedure: Bronchoalveolar Lavage
- Group C (Experimental): Bronchoalveolar lavage with acetylcysteine solution in combination with saline on the basis of conventional clinical treatment, with a volume of 90 ml per target lung lobe, up to a maximum of 2 lobes, and a total volume of up to 180 ml.
  Interventions: Procedure: Bronchoalveolar Lavage

INTERVENTIONS:
Procedure: Bronchoalveolar Lavage — Bronchoalveolar lavage with saline or saline-acetylcysteine solution on the basis of conventional clinical treatment, with a volume of 90 ml per target lung lobe, up to a maximum of 2 lobes, and a total volume of up to 180 ml.
  Arms: Group B; Group C

SUMMARY:
Bronchiectasis is a clinical syndrome characterised by chronic cough, profuse sputum and/or intermittent haemoptysis, with or without shortness of breath and respiratory failure of varying severity, and abnormal thickening and dilatation of the bronchial walls as seen on lung imaging. Nebulised inhalation of N-acetylcysteine has been shown to significantly improve symptoms, shorten the length of hospital stay, reduce the rate of re-hospitalisation within six months, and improve lung function in patients with bronchiectasis with a high degree of safety. There have been no studies on the efficacy and safety of bronchoscopic irrigation with N-acetylcysteine solution in the treatment of bronchiectasis. The aim of this study was to investigate whether bronchoscopic acetylcysteine lavage combined with conventional treatment is more beneficial to patients with bronchiectasis than conventional treatment combined with conventional bronchoalveolar lavage and conventional treatment without bronchoscopy, respectively.

DETAILED DESCRIPTION:
All patients enrolled were patients with acute exacerbation of bronchiectasis. A total of 180 patients (1:1:1 allocation) with acute exacerbation of bronchiectasis were to be enrolled. The patients were divided into control group A (conventional clinical treatment including anti-infective and expectorant therapy), control group B (bronchoalveolar lavage with saline on the basis of conventional clinical treatment, with a volume of 90 ml per target lung lobe, up to a maximum of 2 lobes, and a total volume of up to 180 ml), and experimental group C (bronchoalveolar lavage with acetylcysteine solution in combination with saline on the basis of conventional clinical treatment, with a volume of 90 ml per target lung lobe, up to a maximum of 2 lobes, and a total volume of up to 180 ml).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80 years;
2. Chest CT suggestive of bronchiectasis;
3. meet the criteria for an acute exacerbation of bronchiectasis with symptoms such as cough, sputum, chest tightness or wheezing, and c. Patients who meet the criteria for an acute exacerbation of bronchiectasis with symptoms of cough, sputum, chest tightness or wheezing and who consent to bronchoscopy with bronchoalveolar lavage
4. patients who agreed to participate in the study and signed an informed consent form;

Exclusion Criteria:

1. Severe cardiopulmonary diseases, coagulation disorders, poor tolerance to anaesthesia, psychiatric disorders or severe neuroses that are contraindications to bronchoscopy;
2. Intraoperative findings of decreased SPO2 or inability to tolerate bronchoscopy or inability to tolerate further bronchoalveolar lavage;
3. Inability to co-operate with the study for any reason or in the opinion of the investigator, inappropriate for inclusion in the study for other reasons;
4. Bronchoscopy of patients with significant intra-airway haemorrhage who may be at risk of exacerbation due to bronchoalveolar lavage;
5. Patients with acetylcysteine allergy;
6. Missing information;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Time of first and second acute exacerbation | six months
  Description: Length of post-treatment time points to first acute exacerbation (days) and length of time points to second acute exacerbation (days) in all three groups of patients.

SECONDARY OUTCOMES:
The change of mMRC scores | one month
  The modified Medical Research Council (mMRC) of all patients followed up at different time points (day 0, day 3, day 7, one month after treatment). Categorised on a scale of 0 to 4, the higher the scale the more severe the symptoms are.
The change of CAT scores. | one month
  COPD assessment test (CAT) of all patients followed up at different time points (day 0, day 3, day 7, one month after treatment). A score of 0-10 is considered mild, 11-20 is considered moderate, 21-30 is considered severe, and 31-40 is considered very severe.
The change of LCQ scores. | one month
  Leicester Cough Questionnaire (LCQ) of all patients followed up at different time points (day 0, day 3, day 7, one month after treatment). Scores range from 3 to 21, with lower scores suggesting that cough has a greater impact on quality of life.
The change of SGQR scores. | one month
  St George's Respiratory Questionnaire (SGRQ) of all patients followed up at different time points (day 0, day 3, day 7, one month after treatment). The total score ranges from 0 to 100. Higher scores indicate poorer quality of life for the patient.
Number of acute exacerbations | six months
  Number of acute exacerbations in the three groups at 6 months after treatment.
adverse effects | one month
  Occurrence of post-treatment adverse effects (chest tightness, shortness of breath, worsening of respiratory failure, worsening of haemoptysis, complication of new pneumonia foci or signs of significant new infections considered to be related to lavage treatment) in the three groups of patients.
Re-treatment with bronchoalveolar lavage | six months
  Hospitalisation for acute exacerbations requiring re-bronchoscopic lavage within 6 months in all three groups (re-bronchoscopic lavage may be considered for exacerbations after treatment: significant increase in sputum output, increase in the size of the lesion on CT).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No